CLINICAL TRIAL: NCT05392231
Title: Assessment of Fetal Pancreatic Size and Maternal Serum Biomarkers Glycated Albumin and Insulin-regulated Aminopeptidase in Women With Gestational Diabetes Mellitus
Brief Title: Assessment of Fetal Pancreatic Size and Maternal Serum Biomarkers in GDM
Acronym: PS-GDM-2022
Status: Completed | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 05-2022
Record Dates: First submitted 2022-05-22; First posted 2022-05-26 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators aimed to determine the predictive values of fetal pancreas size and maternal serum biomarkers glycated albumin (GA) and insulin-regulated aminopeptidase (IRAP) for gestational diabetes mellitus (GDM).

DETAILED DESCRIPTION:
The investigators aimed to determine the predictive values of fetal pancreas size and maternal serum biomarkers glycated albumin (GA) and insulin-regulated aminopeptidase (IRAP) for gestational diabetes mellitus (GDM).In this prospective observational study including 109 pregnant women, the fetal pancreas size and maternal serum biomarkers GA and IRAP were measured at the gestational age of 20-22 weeks and later at the gestational age of 24-28 weeks, in 19 participants of them, GDM was confirmed with the 75-g oral glucose tolerance test (OGTT) and the fetal pancreas size was measured in all the participants again.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age between 18 and 42 years
* Gestational age between 20 and 28 weeks

Exclusion Criteria:

* Multiple pregnancies
* Pregestational diabetes
* Fetal congenital malformations
* Placental and amniotic fluid abnormalities
* Preeclampsia
* Severe systemic disease
* Long-term systemic drug usage

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: With a design of prospective observational study, this research was carried out in the Perinatology Clinic of Haseki Hospital, affiliated with the University of Health Sciences, in Istanbul, between September 2021 and April 2022, following the approval of the local ethics committee (date: February 09, 2022, Registry No: 05-2022) and the valid Helsinki Declaration. After all the objectives of this work and context of all the procedures that could be undertaken were properly explained to each pregnant woman, the participant was requested to sign an informed written consent form.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Early prediction of gestational diabetes | Two months
  Early prediction of gestational diabetes by the fetal pancreas measurement with ultrasound and maternal serum biomarkers glycated albumin and insulin-regulated aminopeptidase measured with ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Guleroglu FY, Ozmen AB, Bakirci IT, Dogu SY, Yilmaz I, Cetin A. Fetal pancreas size and maternal serum biomarkers glycated albumin and insulin-regulated aminopeptidase provide no potential for early prediction of gestational diabetes mellitus. Arch Gynecol Obstet. 2023 Nov;308(5):1505-1514. doi: 10.1007/s00404-022-06860-2. Epub 2022 Nov 27. PMID 36436013